CLINICAL TRIAL: NCT01783756
Title: Phase 1b/2 Single-arm Trial Evaluating the Combination of Lapatinib, Everolimus and Capecitabine for the Treatment of Patients With HER2-positive Metastatic Breast Cancer With CNS Progression After Trastuzumab
Brief Title: Phase 1b/2 Trial Using Lapatinib, Everolimus and Capecitabine for Treatment of HER-2 Positive Breast Cancer With CNS Metastasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRIO-US B09; NCI-2013-00082 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 12-001358 (Other: UCLA IRB)
Record Dates: First submitted 2013-01-31; First posted 2013-02-05 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Central Nervous System Metastases; HER2-positive Breast Cancer; Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine; Everolimus; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (lapatinib ditosylate, everolimus, capecitabine) (Experimental): Patients receive lapatinib ditosylate PO QD and everolimus PO QD on days 1-21, and capecitabine PO BID on days 1-14. Treatment repeats every 21 days for 17 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lapatinib ditosylate; Drug: everolimus; Drug: capecitabine; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lapatinib ditosylate — Given PO
  Other Names: GSK572016; GW-572016; GW2016; Lapatinib; Tykerb
Drug: everolimus — Given PO
  Other Names: 42-O-(2-hydroxy)ethyl rapamycin; Afinitor; RAD001
Drug: capecitabine — Given PO
  Other Names: CAPE; Ro 09-1978/000; Xeloda
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This is a phase 1b/2 study to evaluate the safety and clinical activity of the combination of lapatinib, everolimus and capecitabine for the treatment of participants with HER2+ breast cancer with metastases in the brain who have progressed on trastuzumab.

The combination of 2 drugs able to reach the brain (lapatinib and everolimus) that target different parts of the HER2 signaling pathway plus chemotherapy (capecitabine) that has proven benefits in metastatic breast cancer may lead to improved clinical outcomes for participants with CNS metastasis.

Participants will undergo brain MRIs and CT scans of the chest and abdomen to evaluate response to the treatment, regular laboratory tests and echocardiogram or Multi Gated Acquisition Scan (MUGA) to assess cardiac activity

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Central nervous system (CNS) objective response rate at 12 weeks: defined as either a complete response or partial response provided there is no progression of extra-CNS disease, increasing steroid requirements, or worsening of neurologic signs and symptoms (NSS)^34 Lesions will be measured using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

SECONDARY OBJECTIVES:

I. Safety and tolerability. II. Median progression free survival. III. Median overall survival. IV. CNS objective response rate and clinical benefit rate (complete response, partial response and stable disease lasting at least 6 months).

V. Extra-CNS objective response rate according to RECIST1.1.

OUTLINE:

Patients receive lapatinib ditosylate orally (PO) once daily (QD) and everolimus PO QD on days 1-21, and capecitabine PO twice daily (BID) on days 1-14. Treatment repeats every 21 days for 17 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment or treatment discontinuation, patients will complete 2 follow up visits within 7 days and at 30 days and then will be followed for survival every 3 months for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HER2+ (immunohistochemistry [IHC] 3+ or fluorescence in situ hybridization [FISH]+ R/G > 2.0 or silver-enhanced in situ hybridization [SISH]+ HER2/chromosome 17 centromere [CEP17] > 2.0) breast cancer with documented central nervous system (CNS) recurrence or progression
* Must have received trastuzumab (neoadjuvant, adjuvant or metastatic setting)
* At least one measurable lesion in the brain (>= 10 mm on T1-weighted, gadolinium-enhanced magnetic resonance imaging [MRI]); (prior neurosurgical resection, whole brain radiation or stereotactic radiation therapy is allowed provided the patient has a measurable CNS progression [at least one new and/or progressive measurable brain metastasis]; measurable or non-measurable extracranial metastases allowed)
* Concurrent steroids allowed (up to equivalent of prednisone 20 mg daily, on taper or stable dose for at least 2 weeks)
* Life expectancy of >= 12 weeks
* Previous treatment with other HER2 targeted agents allowed; (previous treatment with HER2 inhibitors and investigational drugs to be discontinued prior to starting study treatment [at least 21 days for trastuzumab and other antibodies; at least 14 days for lapatinib; at least 5 half-lives for other agents])
* Previous chemotherapy (adjuvant and metastatic regimens) and hormonal therapy allowed, but chemotherapy must have been discontinued at least 21 days prior to starting study treatment and hormonal therapy at least 7 days prior to starting study treatment; patients must have recovered from acute Common Terminology Criteria for Adverse Events (CTCAE) v 4.0 grade >= 2 side effects of previous treatments
* At least 2 weeks since prior radiotherapy or stereotactic radiosurgery, and 4 weeks since prior major surgery at time of study enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin (Hb) >= 9 g/dL
* Serum bilirubin =< 1.5 x upper limit of normal (ULN) (=< 3.0 if Gilbert's syndrome)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN (=< 5 x ULN in patients with liver metastases)
* International normalized ratio (INR) =< 1.5
* Adequate renal function: serum creatinine =< 1.5 x ULN
* Fasting serum cholesterol =< 300 mg/dL OR =< 7.75 mmol/L AND fasting triglycerides =< 2.5 x ULN; NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication
* Signed informed consent
* Age >= 18 years

Exclusion Criteria:

* Patients who have never received trastuzumab
* Prior treatment with an mammalian target of rapamycin (MTOR) inhibitor (including everolimus, sirolimus, temsirolimus)
* Leptomeningeal carcinomatosis as only site of CNS disease
* Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Patients with clinically significant interstitial lung disease or history of cardiac disease
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study
* Prior treatment with any investigational drug within the preceding 4 weeks prior to starting study drug
* Patients receiving chronic, systemic treatment with corticosteroids (more than 20 mg/day prednisone equivalent, see inclusion criteria) or another immunosuppressive agent; topical or inhaled corticosteroids are allowed
* Patients should not receive immunization with attenuated live vaccines within one week of starting study drug or during study period; close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus; examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, Bacillus Calmette-Guérin (BCG), yellow fever, varicella and typhoid vaccine live oral (TY)21a typhoid vaccines
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * Symptomatic congestive heart failure of New York heart Association class III or IV
  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia, left ventricular ejection fraction (LVEF) < 50% or any other clinically significant cardiac disease
  * Severely impaired lung function as defined as spirometry and diffusion capacity of the lung of carbon monoxide (DLCO) that is 50% of the normal predicted value and/or oxygen (02) saturation that is 88% or less at rest on room air
  * Uncontrolled diabetes as defined by fasting serum glucose > 1.5 x ULN (Note: optimal glycemic control should be achieved before starting trial therapy)
  * Active (acute or chronic) or uncontrolled severe infections
  * Liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C)
  * Note: A detailed assessment of hepatitis B/C medical history and risk factors must be done at screening for all patients; hepatitis B virus (HBV) deoxyribonucleic acid (DNA) and hepatitis C ribonucleic acid polymerase chain reaction (HCV RNA PCR) testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection; patients with positive results for HBV/HCV infection will be allowed in this study provided monitoring and prophylactic treatment are followed
* A known history of human immunodeficiency virus (HIV) seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus/lapatinib (lapatinib ditosylate) (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active, bleeding diathesis
* Patients on warfarin (patients on injectable blood thinners, such as Lovenox, are able to continue those)
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods; adequate contraception must be used throughout the trial and for 8 weeks after the last dose of study drug, by both sexes; (women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of study drug)
* Male patient whose sexual partner(s) are women of childbearing potential (WOCBP) who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment
* Patients with a known hypersensitivity to everolimus or other rapamycins (e.g., sirolimus, temsirolimus) or to its excipients
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-06-26; Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
CNS objective response rate defined as either a complete response or partial response provided there is no progression of extra-CNS disease, increasing steroid requirements, or worsening of NSS measured using RECIST v1.1 | 12 weeks
  Estimated with a 95% confidence interval. Chi-square test will be used evaluate if the CNS response rate at week 12 is significantly higher than 20%.

SECONDARY OUTCOMES:
Body system, severity and relation with study treatment of adverse events graded according to the National Institute of Health (NIH)/ National Cancer Institute (NCI) Common Toxicity Criteria (CTC) v4.0 | Up to 12 months
Progression-free survival (PFS) by the RECIST v1.1 | Interval between the date of study enrollment and the earliest date of disease progression, assessed up to 1 year after end of treatment
  The distribution of PFS and OS will be estimated using Kaplan-Meier method and survival curves for PFS and OS will be plotted. Median PFS and median OS will be obtained.
Overall survival (OS) | Interval between the date of study enrollment and the date of death, assessed up to 12 months after end of treatment
  The distribution of PFS and OS will be estimated using Kaplan-Meier method and survival curves for PFS and OS will be plotted. Median PFS and median OS will be obtained.
Extra CNS response according to RECIST1.1 | 12 weeks
  Will be analyzed similarly to CNS objective response rate.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Hurvitz, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Hurvitz S, Singh R, Adams B, Taguchi JA, Chan D, Dichmann RA, Castrellon A, Hu E, Berkowitz J, Mani A, DiCarlo B, Callahan R, Smalberg I, Wang X, Meglar I, Martinez D, Hobbs E, Slamon DJ. Phase Ib/II single-arm trial evaluating the combination of everolimus, lapatinib and capecitabine for the treatment of HER2-positive breast cancer with brain metastases (TRIO-US B-09). Ther Adv Med Oncol. 2018 Nov 9;10:1758835918807339. doi: 10.1177/1758835918807339. eCollection 2018. PMID 30542377